CLINICAL TRIAL: NCT00694135
Title: A Prospective, Multi-Center, Randomized, Double-Masked, Safety, Tolerability and Efficacy Study of Four Iontophoretic Doses of Dexamethasone Phosphate Ophthalmic Solution in Patients With Non-Infectious Anterior Segment Uveitis
Brief Title: Safety and Efficacy Study of Iontophoresis and Dexamethasone Phosphate to Treat Anterior Uveitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eyegate Pharmaceuticals, Inc. (Industry)
Responsible Party: Stephen From, President and Chief Executive Officer, Eyegate Pharmaceuticals, Inc.
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EGP-437-001
Record Dates: First submitted 2008-06-05; First posted 2008-06-10 (Estimated); Last update posted 2010-08-31 (Estimated); Status verified 2010-08

CONDITIONS: Uveitis, Anterior
Keywords: Iontophoresis; Non-Infectious Acute Anterior Segment Uveitis; Ophthalmology
MeSH Terms: conditions — Uveitis, Anterior

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- EGP-437 1.6 mA-min at 0.4 mA (Active Comparator): Ocular iontophoresis with EGP 437 1.6 mA-min at 0.4 mA
  Interventions: Drug: EGP-437 1.6 mA-min at 0.4 with EyeGate® II System
- EGP-437 4.8 mA-min at 1.2 mA (Active Comparator): Ocular iontophoresis with EGP-437 4.8 mA-min at 1.2 mA
  Interventions: Drug: EGP-437 4.8 mA-min at 1.2 mA with EyeGate® II System
- EGP-437 10.0 mA-min at 2.5 mA (Active Comparator): Ocular iontophoresis with EGP-437 10.0 mA-min at 2.5 mA
  Interventions: Drug: EGP-437 10.0 mA-min at 2.5 mA with EyeGate® II System
- EGP-437 14.0 mA-min at 3.5 mA (Active Comparator): Ocular iontophoresis with EGP-437 14.0 mA-min at 3.5 mA
  Interventions: Drug: EGP-437 14.0 mA-min at 3.5 mA with EyeGate® II System

INTERVENTIONS:
Drug: EGP-437 1.6 mA-min at 0.4 with EyeGate® II System — Ocular Iontophoresis with EGP-437 1.6 mA-min at 0.4 mA delivered via EyeGate® II Drug Delivery System
  Other Names: Dexamethasone Phosphate Ophthalmic Solution
  Arms: EGP-437 1.6 mA-min at 0.4 mA
Drug: EGP-437 4.8 mA-min at 1.2 mA with EyeGate® II System — Ocular Iontophoresis with EGP-437 4.8 mA-min at 1.2 mA delivered via EyeGate® II Drug Delivery System
  Other Names: Dexamethasone Phosphate Ophthalmic Solution
  Arms: EGP-437 4.8 mA-min at 1.2 mA
Drug: EGP-437 10.0 mA-min at 2.5 mA with EyeGate® II System — Ocular Iontophoresis with EGP-437 10.0 mA-min at 2.5 mA delivered via EyeGate® II Drug Delivery System
  Other Names: Dexamethasone Phosphate Ophthalmic Solution
  Arms: EGP-437 10.0 mA-min at 2.5 mA
Drug: EGP-437 14.0 mA-min at 3.5 mA with EyeGate® II System — Ocular Iontophoresis with EGP-437 14.0 mA-min at 3.5 mA delivered via EyeGate® II Drug Delivery System
  Other Names: Dexamethasone Phosphate Ophthalmic Solution
  Arms: EGP-437 14.0 mA-min at 3.5 mA

SUMMARY:
The purpose of this study is to define a safe and effective dose of iontophoretic delivery of dexamethasone phosphate ophthalmic solution using the EyeGate® II Drug Delivery System in patients with non-infectious anterior segment uveitis.

DETAILED DESCRIPTION:
This is a randomized, double-masked, parallel group, dose-comparison, exploratory study of four doses of iontophoretic delivery of dexamethasone phosphate ophthalmic solution in patients with non-infectious anterior segment uveitis. The current study will evaluate the safety, tolerability, and efficacy of this technology at the four dose levels to determine a safe effective dose appropriate for future trials.

ELIGIBILITY:
Inclusion Criteria:

• Non-infectious anterior uveitis

Exclusion Criteria:

* Uveitis of infectious etiology
* Previous anterior uveitis episode ≤ 4 weeks prior to baseline
* Intraocular pressure (IOP) ≥ 25 mmHg at baseline, a history of glaucoma, and/or patients who require ocular anti-hypertensive medications
* Topical corticosteroid treatment in either eye < 48 hours prior to baseline
* Oral corticosteroid or intraorbital corticosteroid treatment in either eye < 2 weeks prior to baseline
* Active intermediate or posterior uveitis

Ages: 12 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2008-06; Primary Completion 2009-07 (Actual); Study Completion 2009-08 (Actual)

PRIMARY OUTCOMES:
Proportion of subjects with an ACC score of zero at Days 14 and 28 | Prospective study, subjects followed for 28 days
  Proportion of subjects with an anterior chamber cell (ACC) score of zero at Days 14 and 28

SECONDARY OUTCOMES:
Time to ACC score of zero | Prospective study, subjects followed for 28 days
  Time to anterior chamber cell score of zero
Proportion of subjects with a reduction of one full ACC score or more from baseline at Day 28 | Prospective study, subjects followed for 28 days
  Proportion of subjects with a reduction of one full anterior chamber cell score or more (≥ 0.5 decrease) from baseline at Day 28
Change from baseline in ACC score at Day 28 | Prospective study, subjects followed for 28 days
  Change from baseline in anterior chamber cell score at Day 28
Treatment emergent adverse events | Prospective study, subjects followed for 28 days
  Treatment emergent adverse events

CONTACTS AND LOCATIONS:
Overall Officials: C. Stephen Foster, MD, Principal Investigator — Massachusetts Eye Research and Surgery Institution; Michael Raizman, MD, Principal Investigator — Ophthalmic Consultants of Boston
Locations (19):
- United States (13):
  - University of Miami, Miami, Florida
  - Emory Eye Center, Atlanta, Georgia
  - Ophthalmic Consultants of Boston, Boston, Massachusetts
  - Massachusetts Eye Research and Surgery Institution, Cambridge, Massachusetts
  - Comprehensive Eye Care Ltd., Washington, Missouri
  - New York Eye & Ear Infirmary, New York, New York
  - Cleveland Eye Clinic, Cleveland, Ohio
  - Oregon Health Services University, Portland, Oregon
  - Pennsylvania College of Optometry, Elkins Park, Pennsylvania
  - Scheie Eye Institue, Philadelphia, Pennsylvania
  - Southern College of Optometry, Memphis, Tennessee
  - Texas Retina Associates, Dallas, Texas
  - Virginia Eye Consultants, Norfolk, Virginia
- India (6):
  - St. Johns Medical College and Hospital, Bangalore, Karnataka
  - Vittala International Institute of Ophthalmology, Bangalore, Karnataka
  - Narayana Nethralaya, Bangalore, Karnataka
  - M. M. Joshi Eye Institute, Hubli, Karnataka
  - Kasturba Medical College and Hospital, Manipal, Karnataka
  - Christian Medical College, Vellore, Tamil Nadu